CLINICAL TRIAL: NCT02340689
Title: Genetic Characterization and Genotype/Phenotype Correlations in Primary Hyperoxaluria
Brief Title: Primary Hyperoxaluria Mutation Genotyping/Phenotyping
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, Principal Investigator, Mayo Clinic
Other Study IDs: 13-006384
Record Dates: First submitted 2014-09-16; First posted 2015-01-19 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Primary Hyperoxaluria
Keywords: PH; PH type 1; Primary Hyperoxaluria; Hyperoxaluria; Primary Oxalosis; PH type 2; PH type 3; Genetic testing for PH; Genetic testing for Primary Hyperoxaluria; Hereditary study for PH; Hereditary study for Primary Hyperoxaluria; AGXT; GRHPR; HOGA1
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria | interventions — Genetic Testing; Hydrogen-Ion Concentration; serine-pyruvate aminotransferase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples retained for potential future use, with consent of subjects only.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Genetic testing: Genetic Analysis
  Interventions: Other: Genetic Analysis

INTERVENTIONS:
Other: Genetic Analysis — We will draw one tube of blood from your arm to obtain white blood cells. These white blood cells will be used as a source of DNA for genetic analysis.
  Other Names: PH; PH type 1; Primary Hyperoxaluria; Hyperoxlauria; Primary Oxalosis; PH type 2; PH type 3; Genetic testing for PH; Genetic testing for Primary Hyperoxaluria; Hereditary study for PH; Hereditary study for Primary Hyperoxaluria; AGXT; GRHPR; HOGA1

SUMMARY:
Specific mutations relating to hyperoxaluria will be determined via DNA analysis by the Mayo RKSC research staff.

DETAILED DESCRIPTION:
During your study visit, we will draw one tube, about two teaspoons (1 to 1 ½ teaspoons for children), of blood from your arm. White blood cells from the sample will be used as a source of DNA for genetic testing. We will use the DNA to try to identify mutations (changes) in one of the genes that can cause primary hyperoxaluria. This will be done by comparing it with the structure of these genes in normal individuals, patients with primary hyperoxaluria, and family members of primary hyperoxaluria patients. In family members of primary hyperoxaluria patients, a 24 hr urine test may also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Ages birth to 99 years in whom clinical information is available from medical records
* Patients with a diagnosis of PH confirmed on previous genetic testing
* Patients with clinical suspicion of primary hyperoxaluria (elevated urine oxalate of greater than 0.8 mmol/1.73 m2/day (>70 mg/1.73 m2/day), history of kidney stones, and/or nephrocalcinosis documented by medical history or imaging studies
* First or second degree family members of a patient with primary hyperoxaluria

Exclusion Criteria:

* Stone formers who do not have confirmed PH and do not meet the inclusion criteria for clinical suspicion of primary hyperoxaluria
* Unwilling or unable to provide consent/assent.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with clinical characteristics suggesting of primary hyperoxaluria
  * Family members of patients with clinical characteristics suggestive of primary hyperoxaluria
Sampling Method: Non-Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Genotype markers of early symptomatic onset of primary hyperoxaluria | 5 years
  Correlation of genotype with severity of disease as defined by age at onset of symptoms

SECONDARY OUTCOMES:
Genotype markers of marked hyperoxaluria in patients with primary hyperoxaluria | 5 years
  Correlation of genotype with severity of disease as defined by the level of urine oxalate
Genotype markers of early loss of kidney function in patients with primary hyperoxaluria. | 5 years
  Correlation of genotype with age at kidney failure

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Milliner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Using a limited data set, plans to share data in accordance with NIH funding expectations.

REFERENCES:
- See also: Mayo Clinic Hyperoxaluria Center — http://www.mayoclinic.org/nephrology-rst/hyperoxaluriacenter.html
- See also: Mayo Clinic Hyperoxaluria and Oxalosis — http://www.mayoclinic.org/hyperoxaluria